CLINICAL TRIAL: NCT01793480
Title: Phase IIIb Evaluation of the Efficacy and Safety of Two Methadone Titration Methods for the Treatment of Cancer-related Pain With Inadequate Pain Relief or Intolerable Side Effects When Treated With Level 3 Opioids.
Brief Title: Evaluation of the Efficacy and Safety of Two Methadone Titration Methods for the Treatment of Cancer-related Pain With Inadequate Pain Relief or Intolerable Side Effects When Treated With Level 3 Opioids.
Acronym: EQUIMETH2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-004609-26
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Pain Related to Cancer
Keywords: Methadone in cancer pain
MeSH Terms: interventions — Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patient-controlled dose of methadone (Experimental): The titration will be done on the patient's request (patient-controlled dose of methadone), with no overlapping with the previous opioid treatment, under the investigator's supervision.
  Interventions: Drug: Methadone
- fixed-dose of methadone (Experimental): The titration will be done with fixed-dose of methadone, on a progressive switch with overlapping with the previous opioid treatment, to avoid withdrawal syndrome when the opioid is discontinued.
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone

SUMMARY:
This is a multicentric, randomized, open-label, phase IIIb national study, to evaluate the clinical effects (success/failure) of methadone for the treatment of cancer-related-pain in patients with inadequate pain relief or intolerable side effects when treated with level 3 opioid.

Principal objective is to compare the clinical effects (success/failure) of two methods of methadone titration in patients with cancer-related pain inadequately relieved or with intolerable side effects after treatment with level 3 opioid.

Secondary objectives are : Overall safety of methadone during the study, to describe the patients' characteristics, to describe the effects of methadone on pain relief, to describe the methadone administration, to evaluate patient's quality of life, to evaluate the prescriber's opinion regarding the handling of methadone initiation.

DETAILED DESCRIPTION:
The randomisation (1:1) will consider the two titration methadone switching methods:

* Group A: patient-controlled dose of methadone with no overlapping with the previous opioid treatment
* Group B: fixed-dose of methadone with overlapping with the previous opioid treatment

Study Description:

Screening visit (Visit 1) within 48 hours before the inclusion Inclusion visit (Visit2) and randomisation on Day 1 Visit 3 from Day 2 to Day 7 (hospitalisation for all patients). Four follow-up visits on Day 14 (Visit 4), Day 21(Visit 5), Day 28 (Visit 6), Day 42 (Visit 7) End of study visit on Day 56 Follow-up phone contact on Day 84.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient of at least 18 years of age
* Patient suffering from cancer disease, undergoing chemotherapy treatment or not, hospitalised or requiring hospitalisation
* Patient presenting nociceptive or mixed pains inadequately relieved with level 3 opioids (morphine, oxycodone, transdermal fentanyl, hydromorphone) with a numeric pain scale score ≥5 evidence-based or presenting intolerable side effects with level 3 opioids
* Patient undergoing level 3 opioid treatment (morphine sulphate or morphine chlorhydrate or fentanyl or oxycodone or hydromorphone)
* Patient presenting a good understanding of the study objectives and able to give his/her written consent
* Patient able to communicate with the investigator or his representative
* Patient available during the whole course of the study and agreeing the study requirements
* Patient with Social Insurance
* Patient having received patient's information form, orally informed and having signed the consent form

Exclusion Criteria:

* Patient in terminal cancer disease (life expectancy less than 2 months) according to investigator's judgement
* Patient treated with a medication that may result in an interaction with methadone, such as: antiarrythmic treatments (Ia or III), erythromycin, spiramycin, intravenous vincamin
* Patient receiving opioid treatment for any other reason than pain
* Patient unable to swallow the study treatment
* Patient presenting contra-indication to the use of methadone
* Patient having a decompensated respiratory failure or a severe hepatic disease
* Patient having a known hypersensitivity to methadone
* Patient presenting QT interval prolongation on ECG results
* Patient receiving a concomitant treatment with a morphine-type agonist-antagonist medication (pentazocine, buprenorphine, nalbuphine) or with sultopride, or with morphinic antagonist (naltrexone)
* Patient treated by analgesic radiotherapy within 15 days before inclusion
* Patient participating or having participated in another clinical trial with a new therapy within one month before inclusion
* Patient with a history of substance abuse
* For woman with childbearing potential: pregnancy or breastfeeding.
* Forfeiture of freedom or under guardianship
* Past history of suicidal attempts
* Patient likely not to respect the study conditions and/or study discontinuation criteria according to investigator's judgement
* Patient presenting any other medical condition or illness or clinically significant abnormal findings on the physical examination at screening that, in the opinion of the Investigator, make the patient unsuitable for the study or put the patient at additional risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2012-01-05 (Actual); Primary Completion 2014-05-06 (Actual); Study Completion 2014-08-31 (Actual)

PRIMARY OUTCOMES:
Binary main criterion based on success/failure rate related to methadone switch on Day 4. | Day 4
  The success is defined as the adequate pain relief on Day 4 and no occurrence of overdose between Day 1 and Day 4. All unmet definition of success will be considered as a failure.
  The adequate pain relief is defined as the composite criterion:
  * Decrease of at least 2 points on the pain numeric scale from 0 (no pain) to 10 (unacceptable pain) evaluated on Day 4 when compared to the pain numeric scale score at baseline,
  * And a pain numeric scale score <5 during two consecutive days (between Day 1 and Day 4)

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - Investigational Site 10, Amiens
  - Investigational Site 06, Bayonne
  - Investigational Site 13, Caen
  - Investigational Site 03, Gap
  - Investigational Site 11, Le Chesnay
  - Investigational Site 07, Lille
  - Investigational Site 16, Lyon
  - Investigational Site 12, Nice
  - Investigational Site 14, Paris
  - Investigational Site 02, Pierre-Bénite
  - Investigational Site 05, Reims
  - Investigational site 08, Strasbourg
  - Investigational Site 17, Suresnes
  - Investigational Site 01, Tarbes
  - Investigational Site 04, Toulouse
  - Investigational Site 15, Villejuif